CLINICAL TRIAL: NCT04629625
Title: The Effect of End-range Mobilization on Time Curve of Pressure Pain Threshold in Knee Osteoarthritis
Brief Title: End-range Mobilization on Time Curve of Pressure Pain Threshold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pecs (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MaitlandKneePPT_Time Curve
Record Dates: First submitted 2020-10-28; First posted 2020-11-16 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Knee Osteoarthritis
Keywords: Musculoskeletal Manipulations; Osteoarthritis, Knee; Pain Threshold
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- End-range mobilization (Experimental): End-range mobilization performed in end-position of the tibiofemoral joints' flexion and extension for 2*3 min
  Interventions: Biological: End-range mobilization
- Non end-range mobilization (Active Comparator): Non end-range mobilization performed in tibiofemoral joints' loose position
  Interventions: Biological: Non end-range mobilization
- Placebo (Placebo Comparator): Hands-on treatment technique performed in end-range of the tibiofemoral joints' flexion and extension for 2*3 min
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: End-range mobilization — End-range mobilization performed in end-range of the tibiofemoral joints' flexion and extension
  Arms: End-range mobilization
Biological: Non end-range mobilization — Non end-range mobilization performed in tibiofemoral joints' loose position
  Arms: Non end-range mobilization
Biological: Placebo — Hands-on technique performed in end-range of the tibiofemoral joints' flexion and extension
  Arms: Placebo

SUMMARY:
Pain in knee osteoarthritis (OA) represents increased pain intensity due to peripheral and central sensitivity. Pressure pain threshold (PPT) is a widely applied technique for measuring the magnitude of peripheral and central sensitivity in knee OA. Despite several manual therapy techniques has been proven to increase PPT in knee OA, the effect of end-range mobilization on the time curve of PPT has not been evaluated so far in knee OA. The aim of this study was to investigate the effect of end-range mobilization on the time curve of PPT and some function-related measures in knee OA.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is the most common form of arthritis leading to a major disability worldwide. Although many mechanisms may contribute to knee pain severity, the patient-reported hyperalgesia can be attributed to peripheral and central sensitivity in knee OA. Amongst quantitative sensory testing methods, pressure pain threshold (PPT) measurement is a simple and commonly applied method for measuring somatosensory function in musculoskeletal disorders, just as in knee OA. Many trials have presented lower PPT in knee OA compared to healthy controls underlining the presence of peripheral and central sensitivity.

The different joint-based mobilization techniques may not only alleviate pain, but also increase pain tolerance to the locally applied mechanical pressure. Positive results of these techniques on increase of PPT has been reported in knee OA; however, the time curve of PPT has not evaluated so far in knee OA. Therefore, the aim of this study was to investigate the effect of end-range mobilization on the time curve of PPT and some function-related measures in knee OA.

ELIGIBILITY:
Inclusion Criteria:

* the clinical classification criteria of knee OA according to the American College of Rheumatology
* Categorization of patients as End Of Range Problem based on manual therapy
* unilateral/bilateral symptomatic tibiofemoral knee osteoarthritis with radiographic evidence of Kellgren-Lawrence scale between 1 and 3
* pain during weight-bearing activities at least within 6 months
* sufficient mental status

Exclusion Criteria:

* acute inflammation of the knee
* class II. obesity (body mass index, BMI>35kg/m2)
* severe degenerative lumbar spine disease (e.g. spondylolisthesis)
* systemic inflammatory arthritic or neurological condition
* physiotherapy/balneotherapy attendance or manual therapy within 3 months
* intraarticular injections in the prior 12 months
* use of walking aids
* contraindication for manual therapy
* complex regional pain syndrome
* cognitive impairment

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2020-10-10 (Actual); Primary Completion 2021-01-02 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
PPT of the knee | 30 minutes
  pressure pain threshold of the knee

SECONDARY OUTCOMES:
PPT of the m. Extensor Carpi Radialis Longus (ECRL) | 30 minutes
  pressure pain threshold at the ECRL
PPT of the m. Extensor Carpi Radialis Longus (ECRL) | every 2nd day for the following 6-day
  pressure pain threshold at the ECRL
Timed Up and Go test | 30 minutes
  Timed Up and Go test measuring functional capacity
Timed Up and Go test | every 2nd day for the following 6-day
  Timed Up and Go test measuring functional capacity
Strength of passive tension of the knee | 30 minutes
  Strength of passive tension of the knee measured in Newton at the beginning of pain
Strength of passive tension of the knee | every 2nd day for the following 6-day
  Strength of passive tension of the knee measured in Newton at the beginning of pain
Pressure Pain Threshold measurement of the knee | every 2nd day for the following 6-day
  pressure pain threshold measurement of the knee via hand-held algometer

CONTACTS AND LOCATIONS:
Overall Officials: Miklós Pozsgai, Study Chair — Harkány Thermal Rehabilitation Centre
Locations (2):
- Hungary (2):
  - Harkány Thermal Rehabilitation Centre, Harkány, Please Select
  - Miklós Pozsgai, Harkány, Please Select

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kidd BL. Osteoarthritis and joint pain. Pain. 2006 Jul;123(1-2):6-9. doi: 10.1016/j.pain.2006.04.009. Epub 2006 May 22. No abstract available. PMID 16714085
- [Background] Wise BL, Niu J, Zhang Y, Wang N, Jordan JM, Choy E, Hunter DJ. Psychological factors and their relation to osteoarthritis pain. Osteoarthritis Cartilage. 2010 Jul;18(7):883-7. doi: 10.1016/j.joca.2009.11.016. Epub 2010 Mar 24. PMID 20346403
- [Background] Bajaj P, Bajaj P, Graven-Nielsen T, Arendt-Nielsen L. Osteoarthritis and its association with muscle hyperalgesia: an experimental controlled study. Pain. 2001 Aug;93(2):107-114. doi: 10.1016/S0304-3959(01)00300-1. PMID 11427321
- [Background] Imamura M, Imamura ST, Kaziyama HH, Targino RA, Hsing WT, de Souza LP, Cutait MM, Fregni F, Camanho GL. Impact of nervous system hyperalgesia on pain, disability, and quality of life in patients with knee osteoarthritis: a controlled analysis. Arthritis Rheum. 2008 Oct 15;59(10):1424-31. doi: 10.1002/art.24120. PMID 18821657
- [Background] Wylde V, Palmer S, Learmonth ID, Dieppe P. Somatosensory abnormalities in knee OA. Rheumatology (Oxford). 2012 Mar;51(3):535-43. doi: 10.1093/rheumatology/ker343. Epub 2011 Nov 24. PMID 22120461
- [Background] Hendiani JA, Westlund KN, Lawand N, Goel N, Lisse J, McNearney T. Mechanical sensation and pain thresholds in patients with chronic arthropathies. J Pain. 2003 May;4(4):203-11. doi: 10.1016/s1526-5900(03)00557-1. PMID 14622705
- [Background] Kaya Mutlu E, Ercin E, Razak Ozdincler A, Ones N. A comparison of two manual physical therapy approaches and electrotherapy modalities for patients with knee osteoarthritis: A randomized three arm clinical trial. Physiother Theory Pract. 2018 Aug;34(8):600-612. doi: 10.1080/09593985.2018.1423591. Epub 2018 Jan 8. PMID 29308949
- [Background] Khademi-Kalantari K, Mahmoodi Aghdam S, Akbarzadeh Baghban A, Rezayi M, Rahimi A, Naimee S. Effects of non-surgical joint distraction in the treatment of severe knee osteoarthritis. J Bodyw Mov Ther. 2014 Oct;18(4):533-9. doi: 10.1016/j.jbmt.2013.12.001. Epub 2013 Dec 11. PMID 25440203